CLINICAL TRIAL: NCT01530438
Title: Cognitive and Emotional Disorders in Amyotrophic Lateral Sclerosis : Neuropsychological, Imaging and Neuropathological Study
Brief Title: Study of Cognitive and Emotional Disorders in Amyotrophic Lateral Sclerosis
Acronym: SLAMEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 08-067
Record Dates: First submitted 2010-02-22; First posted 2012-02-10 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Magnetic Resonance Spectroscopy

ARMS (3):
- ALS patients without cognitive disorders (Other): Amyotrophic lateral sclerosis without cognitive disorders
  Interventions: Other: MRI + 18FDG-PET + neuropsychological assessments ; 18FDG performed especially for the research
- ALS patients with cognitive disorders (Other): Amyotrophic lateral sclerosis with cognitive disorders
  Interventions: Other: MRI + 18FDG-PET + neuropsychological assessments ; 18FDG performed especially for the research
- ALS patients + frontal-temporal dementia (Other): Amyotrophic lateral sclerosis plus frontal-temporal dementia
  Interventions: Other: MRI + 18FDG-PET + neuropsychological assessments ; 18FDG performed especially for the research

INTERVENTIONS:
Other: MRI + 18FDG-PET + neuropsychological assessments ; 18FDG performed especially for the research — At T0 and T9 or 12 monts, are performed :
  * Imaging : fMRI at rest and anatomical MRI
  * Neuropsychological assessments : general cognitive functioning, theory of mind, executive functions ...

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease that involves not only motor structures, as was previously thought, but also brain areas dealing with cognition as well as parts of the limbic system. Clinical, imaging and pathological evidence suggests that ALS and fronto-temporal dementia (FTD) have several features in common, and that these two diseases could be the two ends of a pathological continuum.

DETAILED DESCRIPTION:
Objectives : the investigators aim to study the clinical profile and magnitude of cognitive disturbances, measure brain metabolism and assess cerebral atrophy in patients with ALS. The relationships between cognitive, metabolic and anatomical data will be determined by the correlation method. In addition, pathological studies will be carried out in deceased patients having given their consent in advance, in order to quantify the neuronal loss and UBIs.

Methods : the investigators plan to recruit 60 patients with ALS, 10 patients with ALS/FTD (the diagnosis of dementia will rest on clinical data and formal neuropsychological testing) and 20 normal control subjects. The ALS patients will be divided into 2 subsets on the basis of a preliminary neuropsychological work-up, according to the presence or absence of "subclinical cognitive impairment" as defined by abnormal scoring on tests not meeting the criteria for dementia. In a second testing session carried out at the same time, a comprehensive assessment of memory, behaviour and emotional changes will be done. All subjects will then undergo morphological magnetic resonance imaging (MRI), resting-state functional MRI and 18-fluorodeoxyglucose positron emission tomography (18FDG-PET). Whenever possible, a second testing session will be carried out 9 to 12 months later in order to quantify the cognitive deterioration, if any, and to find early predictors of the evolution towards dementia. In deceased patients, the location and extent of neuronal loss will be determined, as well as the location and number of UBIs.

Results and clinical relevance : this study is intended to improve our knowledge of the clinical phenotype of ALS, and particularly to learn more about the extent of cognitive, behavioural and emotional changes in this disease. This could in turn shed some further light on the relationships between ALS and FTD.

ELIGIBILITY:
Inclusion Criteria:

* All participants :

  * study level > 7 years
  * mother tongue : french
  * signature of the informed consent of the protocol in accord with the Comité de Protection des Personnes
  * medical, neurological, neuroradiological and neuropsychological approfondis in accord with the specific inclusion and non inclusion criteria spécifiques at each population
* Patients ALS :

  * 18 to 80 years old
  * Diagnostic defined or probable in according to the reviewed criteria of El Escorial.
* Patients ALS / FTD :

  * 18 to 8O years old
  * Diagnostic defined or probable in according to El Escorial reviewed criteria and diagnostic of frontal-temporal dementia in according to Lund et Manchester criteria.
* Control Subjects :

  * 45 to 75 years old
  * DRS ≥ 130
  * BECK < 8

Exclusion Criteria:

* All particpants :

  * Major past history (chronic pulmonary disease, cardiac disease, metabolic, haematological, endocrinological or severe immunological, cancer) ;
  * Chronic use of alcohol or drugs ;
  * IRM contraindications

Protected adults, and persons non affiliated to social protection system won't be able to participate at this study. The inclusion of the participant in another biomedical research protocol(during the study or into 12 months before the inclusion) is too a non inclusion criterion.

* Patients SLA and patients SLA / FTD

  * Severe bulbar disorders
  * Severe restrictive respiratory insufficiency (VC<50%) with orthopny
  * Communication disorders with motor origin (non assessable tests)
* Control Subjects :

  * Pregnant or nursing women
  * Unability to submit at the study medical follow-up for geographic or psychiatric reasons(previous or ongoing).
  * DRS score < 130
  * Depressive syndrome (BECK) ≥ 8

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive, behavioural and emotional changes assesed with Neuropsychological tests. | Between 9 and 12 mth

SECONDARY OUTCOMES:
brain imaging (anatomical MRI, functional MRI, PET using 18FDG) | Between 9 and 12 mth

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Carluer, MD, Principal Investigator — University Hospital, Caen
Locations (2):
- France (2):
  - University Hospital Center, Caen
  - University Hospital Center, Rouen